CLINICAL TRIAL: NCT02713698
Title: Modelling Propofol Pharmacokinetics and Pharmacodynamics During an Intravenous Anaesthesia Guided by the Bispectral Index (BIS)
Brief Title: Propofol Pharmacokinetics and Pharmacodynamics Modelling
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Ana M Araujo, MD, Centro Hospitalar do Porto
Other Study IDs: 2015.221(183-DEFI/165-CES)
Record Dates: First submitted 2016-02-23; First posted 2016-03-21 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Intravenous Anesthetic Agent Overdose
Keywords: Anaesthetics; Intravenous; Propofol; Pharmacokinetics; Pharmacodynamics; Propofol pharmacokinetic-pharmacodynamic model
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood samples will be collected in serum tubes and centrifuged at 2000 rpm for 15 minutes in order to obtain serum. Serum will be preserved at -80ºC until analysis.

GROUPS / COHORTS (3):
- Group 1 (≥18 years, BMI<35kg/m2): Patients with 18 or more years presenting for inpatient nose and ear surgery.
  Interventions: Drug: Propofol
- Group 2 (≥18 years, ≥35kg/m2): Patients with 18 or more years presenting for inpatient bariatric surgery.
  Interventions: Drug: Propofol
- Group 3 (≥65 years): Patients with 65 or more years presenting for orthopaedic surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The whole anaesthetic procedure is standard except for additional body composition assessment with Body Composition Monitor - BCM (Fresenius Medical Care, Germany) and arterial blood samples collection.
  In all included patients, propofol will be started at 2000mg/h until LOC, defined by "loss of eye-lash reflex" and "loss of response to name calling". During surgery propofol infusion will be guided by targeted BIS values between 40 and 60.
  Arterial blood samples will be obtained immediately after LOC and after every 20-30 minutes during propofol infusion. After stopping propofol infusion, arterial blood samples will be acquired every 10 minutes until recovery of consciousness. The maximum blood sample per patient will be 20 mL.

SUMMARY:
The main purpose of this research is to develop a population pharmacokinetic and pharmacodynamic model of Propofol when used for induction and maintenance of anaesthesia, using BIS as a pharmacodynamic endpoint.

A covariate analysis will be performed in order to account for variability in pharmacokinetic and pharmacodynamic parameters. The influence of age and obesity on propofol pharmacokinetic parameters will be particularly addressed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted for nose or ear surgery, bariatric surgery or urgent orthopaedic surgery.

Exclusion Criteria:

* Severe hepatic or renal insufficiency;
* Significant haemodynamic instability previous to the surgery;
* Allergy to eggs or propofol at the time of enrolment;
* Predictive criteria for difficult airway management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient care at Centro Hospitalar do Porto
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

REFERENCES:
- [Derived] Araujo AM, Machado HS, Falcao AC, Soares-da-Silva P. Bioelectrical impedance analysis of body composition for the anesthetic induction dose of propofol in older patients. BMC Anesthesiol. 2019 Oct 11;19(1):180. doi: 10.1186/s12871-019-0856-x. PMID 31604419

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2 (≥18 Years, BMI≥35kg/m2): Patients with 18 or more years presenting for inpatient bariatric surgery.
- Group 3 (≥65 Years): Patients with 65 or more years presenting for urgent orthopaedic surgery.
Period: Overall Study
Arm/Group | Group 1 (≥18 Years, BMI<35kg/m2) | Group 2 (≥18 Years, BMI≥35kg/m2) | Group 3 (≥65 Years)
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (≥18 Years, BMI<35kg/m2) | Group 2 (≥18 Years, BMI≥35kg/m2) | Group 3 (≥65 Years) | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.5) | 47.9 (9.4) | 77.7 (8.6) | 56.4 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 13 | 44
  Male | 7 | 2 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 20 | 20 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Portugal | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Plasma Propofol Concentration (mcg/mL)
Description: Arterial blood samples were obtained after LOC and every 20-30 minutes during propofol infusion. After stopping propofol infusion, arterial blood samples were obtained immediately after recovery of consciousness.
  At the end of the surgery arterial blood samples were centrifuged at 2862xg for 5 minutes and they were preserved at -80ºC until analysis.
  The quantification of propofol in serum was performed using gas chromatography/ion trap-mass spectrometry (GC/IT-MS)
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Group 1 (≥18 Years, BMI<35kg/m2) | Group 2 (≥18 Years, BMI≥35kg/m2) | Group 3 (≥65 Years)
Number analyzed (Participants) | 20 | 20 | 20
mcg/mL | 2.36 (1.38) | 3.12 (1.5) | 2.91 (2.45)

ADVERSE EVENTS:
Time Frame: Perioperative period
Description: The proposed study is a cross sectional analytical study.The whole anaesthetic procedure was standard except for additional body composition assessment with Body Composition Monitor - BCM (Fresenius Medical Care, Germany) and arterial blood samples collection.
Arm/Group | Group 1 (≥18 Years, BMI<35kg/m2) | Group 2 (≥18 Years, BMI≥35kg/m2) | Group 3 (≥65 Years)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (≥18 Years, BMI<35kg/m2) (N=20) | Group 2 (≥18 Years, BMI≥35kg/m2) (N=20) | Group 3 (≥65 Years) (N=20)
Mean arterial pressure (MAP) variation >40% after induction of general anesthesia (Cardiac disorders) | 0 | 1 | 6 — Patients in whom a variation higher than 40% was registered after induction of general anesthesia were treated with ephedrine and fluid boluses to return MAP to baseline levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02713698/Prot_SAP_000.pdf